CLINICAL TRIAL: NCT05422079
Title: Effects of a Motor Control Exercise Protocol Versus a General Exercise Program in Patients With Nonspecific Chronic Low Back Pain: Ultrasound Monitoring
Brief Title: Motor Control Exercises Versus a General Exercise Program in Patients With Nonspecific Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Physiotherapy and Pain Group member, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIM/HU/2019/40
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Low Back Pain
Keywords: Low Back Pain, exercises, ultrasound echography
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single-blind, randomised clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-specific lumbar exercise group (Experimental): Subjects perform a conventional lumbar exercise program twice a week for four weeks.
  Interventions: Other: Non-specific lumbar exercise group
- Group motor control lumbar exercises (Experimental): Subjects perform a lumbar stabilization exercise program twice a week for four weeks.
  Interventions: Other: motor control lumbar exercises
- Group motor control lumbar exercises with ultrasound echography feedack (Experimental): Subjects perform a lumbar stabilization exercise program in conjunction with a video where participants can see how the muscles contract.
  Interventions: Other: motor control lumbar exercises with ultrasound echography feedack

INTERVENTIONS:
Other: Non-specific lumbar exercise group — Subjects perform a conventional lumbar exercise program twice a week.
  Arms: Non-specific lumbar exercise group
Other: motor control lumbar exercises — Subjects perform a lumbar stabilization exercise program.
  Arms: Group motor control lumbar exercises
Other: motor control lumbar exercises with ultrasound echography feedack — Subjects perform a lumbar stabilization exercise program in conjunction with a video where participants can see how the muscles contract.
  Arms: Group motor control lumbar exercises with ultrasound echography feedack

SUMMARY:
The prevalence of low back pain is approximately 49% to 90%, and that 25% of patients seeking treatment for low back pain have a recurrence within the first year. Chronic non-specific low back pain is the most common of all types of pain, not being attributed to a specific pathological cause and with a minimum pain duration of 12 weeks. Forty percent of subjects with acute low back pain will develop chronic low back pain.

Exercise is recommended for the treatment of chronic low back pain because of significant improvements in pain and disability over other therapies, but the evidence is low in the treatment of subacute or acute pain, as exercise appears to be equally effective over rest. Motor control is based on the contraction of the deep and stabilising muscles of the lumbar spine (multifidus and transverse abdominis), performing simple voluntary contraction exercises and increasing (without losing this contraction) their difficulty and functionality. At the beginning, the patient must be able to maintain the isometric contraction of the deep muscles while breathing normally. On the other hand, there is great difficulty in voluntarily contracting the multifidus muscles, especially for subjects with chronic non-specific low back pain, where arthrogenic inhibition hinders their contraction. The application of ultrasound as feedback may help patients to correctly contract this musculature.

Our main objective in the study will be to measure and compare pain, disability, global impression of effect, in patients with non-specific mechanical chronic low back pain after applying a motor control exercise programme with and without ultrasound feedback.

In addition, the investigators will compared this type of exercise with a conventional exercise programme.

DETAILED DESCRIPTION:
A study will be carried out to compare a conventional exercise protocol for the management of non-specific chronic low back pain, with another motor control exercise protocol with and without ultrasound feedback for its correct learning and execution.

For the ultrasound feedback, a video will be recorded where the participant will be able to see how the core muscles contract when each of the motor control exercises is performed.

The participants will be divided into three groups. The first group will perform a general exercise plan for the lower back. The second group will perform a plan of specific motor control exercises aimed at activating the lumbar multifidus and transversus abdominis muscles, and the third group will perform a plan of specific motor control exercises aimed at activating the lumbar multifidus and transversus abdominis muscles using ultrasound as a feedback method.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with low back pain (pain located between the costal margin and the gluteal fold), of non-specific origin, of at least 3 months of evolution.
* Subjects who are not receiving other types of treatment or participating in parallel research.

Exclusion Criteria:

* Muscular diseases that contraindicate the performance of exercise.
* Tumour and/or bone diseases of the dorsolumbar spine.
* Diagnosis of lumbar radiculopathy.
* Women in the process of pregnancy or breastfeeding.
* Consumption of tobacco, alcohol or other substances.
* BMI > 30.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | Change from baseline at 3 months
  This scale assesses the level of pain on a range from 0 to 10, with 0 being no pain and 10 being the maximum possible pain. For a clinically relevant difference to exist, there has to be a difference between measurements of at least 2 points.
  This scale has been shown to have good levels of reliability for pain measurement.

SECONDARY OUTCOMES:
Roland-Morris Disability Questionnarie | Change from baseline at 3 months
  This questionnaire assesses the degree of disability of the patient with low back pain (range 0-24, with 0 being no disability and 24 being total disability). Its Spanish version has been shown to be reliable. To obtain a clinically relevant difference, differences of 1-2 points would be necessary in those patients with low levels of disability, and 7-8 points in those with high levels of disability.
Tampa Scale for Kinesiphobia (TSK-11) | Change from baseline at 3 months
  This questionnaire assesses fear of movement. A minimum detectable change in fear or avoidance behaviour requires 5.6 items. The total score of the scale range from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia, and score ± 37 indicates there is kinesiophobia. This scale has been shown to have an acceptable internal consistency and to be valid.
Patient Global Impression of Change (PGIC) | Change from baseline at 3 months
  The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment. PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."The PGIC is commonly used in clinical studies assessing pain relief following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pecos-Martin, PhD, Study Chair — Alcala University
Locations (2):
- Spain (2):
  - Centro Investigación Fisioterapia y Dolor, Alcalá de Henares, Madrid
  - Physioterapy and Pain center research, Alcalá de Henares, Madrid